CLINICAL TRIAL: NCT01817933
Title: Integrated Rehabilitation Program for Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Ta-Sen Wei,MD, Director, Physical Medical and Rehabilitation, Principal Investigator, Clinical Professor, Changhua Christian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCH-100410
Record Dates: First submitted 2013-03-20; First posted 2013-03-26 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Humeral Neck Fracture; Vertebral Fracture; Distal Radial Fracture; Hip Fractures
MeSH Terms: conditions — Spinal Fractures; Hip Fractures | interventions — Physical Therapy Modalities

ARMS (1):
- Physical therapy (Experimental)
  Interventions: Behavioral: physical therapy

INTERVENTIONS:
Behavioral: physical therapy

SUMMARY:
The recovery of range of motion and muscle power after surgical intervention of the fracture will mostly affect patient's daily activities. So postoperative rehabilitation program will play the important role. Correct and effective physical therapy will reduce the functional impairment of limbs after long term casting or surgical fixation, and accelerate to recover the independent daily activities. There is no consensus between immediate or delay and the duration of continue physical therapy will improve the shoulder function、muscle power and degree of satisfaction( physiological function、social function、mental health、 pain、 general health status ) after surgical fixation of fractures. This study will evaluate the patients of the fracture that including of the humeral neck fracture, vertebral fracture, distal radial fracture and hip fractures after surgical fixation, to see the difference of fracture healing time, function recovery and pain sensation after intervention of physical therapy at different time point.

From this study, we hope to discriminate the timing of intervention and duration of physical therapy which is the key factors for postoperative prognosis of fractures fixation, and to set up the perfect rehabilitation program in ChangHua Christian Hospital. The results of this study will improve the discomfort of fracture patient's recovery or reduce the complications rate, and set up the standard treatment policy of our hospital , also was the model of other hospitals.

ELIGIBILITY:
Inclusion Criteria:

* patients with humeral neck fracture, vertebral fracture, distal radial fracture or hip fractures after surgical fixation

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in pain degree | 1 month after surgical fixation
  use Visual Analog Scale (VAS) to measure the pain condition after surgical fixation and 1 month

SECONDARY OUTCOMES:
Change in range of motion at the fracture area | 1 month after surgical fixation
  to access the range of motion in the elbow, wrist, hip, and knee joint, and the muscle power of upper limb and lower limb